CLINICAL TRIAL: NCT00661154
Title: Avastin/[18-F]-5-fluorouracil PET/CT Imaging Feasibility Project
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GIIMG0001; 97291 (Other: Stanford University Alternate IRB Number); AVF3679s (Other: Genentech)
Record Dates: First submitted 2008-04-14; First posted 2008-04-18 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Colorectal Neoplasms; Colon Cancer; Rectal Cancer; Anal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Anus Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Bevacizumab — 2-12microCi IV injection
  Other Names: Avastin

SUMMARY:
To determine whether using a radiolabelled analog of 5-FU, [18F]-5-fluorouracil, for PET/CT imaging can visually demonstrate differential chemotherapy delivery to known tumor sites before and after administration of bevacizumab and determine the optimal timing of bevacizumab administration to maximize the chemotherapy delivery into the tumor for improved cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed adenocarcinoma of the colon.
2. Patients must have metastatic disease to the liver with at least one lesion that is measurable by RECIST criteria within 4 weeks prior to entry of study
3. Patients with a history of colon adenocarcinoma treated by surgical resection who develop radiological or clinical evidence of metastatic cancer do not require separate histological or cytological confirmation of metastatic disease unless an interval of > 5 years has elapsed between the primary surgery and the development of metastatic disease. Clinicians should consider biopsy of lesions to establish diagnosis of metastatic colon adenocarcinoma if there is substantial clinical ambiguity regarding the nature or source of apparent metastases.
4. Patients must have ECOG performance status of 0-2
5. Patients must be >= 18 years of age
6. Laboratory values <= 2 weeks prior to enrollment:

   * Absolute Neutrophil Count (ANC) >= 1.5 x 10^9/L (>= 1500/mm^3)
   * Platelets (PLT) >= 100 x 10^9/L >= 100,000/mm^3)
   * Hemoglobin (Hgb) >= 9 g/dL
   * Serum creatinine <= 1.5 ULN
   * Serum bilirubin <= 1.5 ULN
   * Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) <= 3.0 x ULN (<= 5 x ULN if liver metastases present). Note: ERCP or percutaneous stenting may be used to normalize the liver function tests.
   * Negative for proteinuria based on dip stick reading OR, if documentation of +1 result for protein on dip stick reading, then total urinary protein <= 500 mg and measured creatinine clearance (CrCl) >= 50 mL/min from a 24-hour urine collection
7. Life expectancy >= 12 weeks
8. Ability to give written informed consent according to local guidelines

Exclusion Criteria:

1. Patients receiving prior 5-FU for the treatment of metastatic colorectal adenocarcinoma will be excluded from enrollment. Previous use of 5-FU for adjuvant treatment of resected stage II or III colorectal adenocarcinoma will be allowed, provided the time from last 5-FU administration to enrollment is > 3 months.
2. Prior full field radiotherapy <= 4 weeks or limited field radiotherapy <= 2 weeks prior to enrollment. Patients must have recovered from all therapy-related toxicities. The site of previous radiotherapy should have evidence of progressive disease if this is the only site of disease.
3. Prior biologic or immunotherapy <= 2 weeks prior to registration. Patients must have recovered from all therapy-related toxicities
4. Prior therapy with anti-VEGF agents
5. Patients with a history of another primary malignancy <= 5 years, with the exception of inactive basal or squamous cell carcinoma of the skin
6. Concurrent use of other investigational agents and patients who have received investigational drugs <= 4 weeks prior to enrollment.
7. Female patients who are pregnant or breast feeding, or adults of reproductive potential not employing an effective method of birth control. Barrier contraceptives must be used throughout the trial in both sexes. Women of childbearing potential must have a negative serum pregnancy test 48 hours prior to administration of study treatment.
8. Patients unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with metastatic (stage IV) colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2008-02; Primary Completion 2009-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Determine whether[18F]-5-Fluorouracil PET/CT scanning can demonstrate a difference in [18F]-5-Fluorouracil tumor uptake before and after the administration of Avastin | 1-4 days

SECONDARY OUTCOMES:
Determine if [18F]-5-Fluorouracil PET/CT imaging demonstrates that there is a difference in maximal [18F]-5-Fluorouracil tumor uptake that is dependent on the time point of post-Avastin scanning | 1-4 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr Andrew Quon, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States